CLINICAL TRIAL: NCT01616394
Title: Postoperative Troponin in Children With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Momeni, MD,PhD; Chef de Clinique Adjointe, Department of Anesthesiology, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: 2011/07/DEC/460
Record Dates: First submitted 2012-02-08; First posted 2012-06-11 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2013-09

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children with congenital heart disease

SUMMARY:
The aim of the study is to evaluate the value of postoperative troponin in the prediction of mid term and long term mortality and morbidity in children with congenital heart disease undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* all children with congenital heart disease between 0-10 years admitted for elective or emergency corrective or palliative cardiac surgery

Exclusion Criteria:

* parental refusal
* children older than 10 years

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with congenital heart disease admitted for surgery
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
mortality | 3 months

SECONDARY OUTCOMES:
morbidity and mortality and length of stay in the PICU and in the hospital | in hospital; 3 months; 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mona MOMENI, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires saint Luc, Brussels, Belgium

REFERENCES:
- [Derived] Momeni M, Poncelet A, Rubay J, Matta A, Veevaete L, Detaille T, Houtekie L, Clement de Clety S, Derycke E, Moniotte S, Sluysmans T, Veyckemans F. Does Postoperative Cardiac Troponin-I Have Any Prognostic Value in Predicting Midterm Mortality After Congenital Cardiac Surgery? J Cardiothorac Vasc Anesth. 2017 Feb;31(1):122-127. doi: 10.1053/j.jvca.2016.02.018. Epub 2016 Feb 23. PMID 27431598